CLINICAL TRIAL: NCT02324205
Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography (ADAPT Trial) ADAPT-BX: Recruitment Plan for Initially Asymptomatic Women Referred for Breast Biopsy
Brief Title: Assessment of Diagnostic Accuracy and Performance of Digital Breast Tomosynthesis Compared to Mammography (ADAPT)
Acronym: ADAPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor met enroll. need for planned second study before meeting enroll. ceiling in protocol
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 124.03-2014-GES-0010_2
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Tumors, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Intervention Model Description: All participants underwent 2D breast imaging with Full-field digital mammography (FFDM) and by 3D breast imaging with Digital Breast Tomosynthesis (DBT).
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBT and FFDM (Experimental): Subjects underwent 2D breast imaging with full-field digital mammography (FFDM) followed by 3D breast imaging with digital breast tomosynthesis (DBT). Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device. Full-Field Digital Mammography: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device.
  Interventions: Device: DBT and FFDM

INTERVENTIONS:
Device: DBT and FFDM — Subjects underwent breast imaging using each device: DBT and FFDM.
  Other Names: Digital Breast Tomosynthesis (3D breast imaging) and Full-Field Digital Mammography (2D breast imaging); 3D breast imaging and 2D breast imaging

SUMMARY:
The aim of this recruitment plan (ADAPT-BX) is to collect image and technical data on both digital breast tomosynthesis (DBT) and full-field digital mammography (FFDM), along with other subject data including histology results from biopsy specimen examination and cancer classification data from initially asymptomatic women referred for biopsy after recall from screening and diagnostic work-up. These data will be included in a subsequent and prospectively planned pooled analysis described in a separate protocol (ADAPT-BIE) examining superiority of DBT to FFDM for breast cancer diagnosis and other clinical performance measures.

DETAILED DESCRIPTION:
ADAPT program consists of 2 recruitment plans (ADAPT-SCR and ADAPT-BX) followed by an off-line read of the images and data collected (ADAPT-BIE). This study involves the comparison of two devices that can identify abnormalities in routine breast screening and diagnostic mammography. Mammography is usually done with full-field digital mammography (FFDM), which takes flat, two-dimensional X-ray images of the breast. Doctors use the two-dimensional images to look for cancers and other abnormal tissue. The purpose of this study is to learn more about the accuracy of full-field digital mammography devices and a new mammography device called digital breast tomosynthesis (DBT). DBT is similar to full-field digital mammography, but can also move around the breast to get X-ray images from different angles, which provides a three-dimensional view that doctors can use to look for cancers and abnormal tissue. Subjects will be recruited from an initially asymptomatic population that have been referred for clinically indicated breast biopsy based on suspicious breast imaging results. Subjects will undergo a DBT mammogram prior to biopsy. If FFDM was not performed within 30 days, subjects will also undergo FFDM prior to biopsy. Results of biopsy(ies) and histopathology, including lesion characteristics, will be recorded and considered as truth if positive for cancer status. Subjects with negative or benign histological findings will be followed for approximately one year (10-16 months) by FFDM and any additional standard of care practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 years or older (≥30 years old);
* Initially asymptomatic women that underwent routine screening FFDM, breast ultrasound (U/S), breast magnetic resonance imaging (MRI) and/or DBT, followed by diagnostic work-up showing one of more abnormalities and referred for breast biopsy within of 30 days before study entry;
* Are able and willing to comply with study procedures;
* Have signed and dated the informed consent form;
* Documented as non-pregnant based on the investigator's medical judgment and in consideration of local clinical practice standards for evidence of non-pregnancy.

Exclusion Criteria:

* Have been previously included in this study;
* Have undergone diagnostic or surgical intervention(s) or procedure(s) on either breast, including mastectomy and cytopunction, before study-related imaging;
* Have breasts too large to be adequately positioned on 24 x 31 centimeter (cm) FFDM digital receptor without anatomical cut off during a DBT examination (or FFDM, if required);
* Have participated in (within the prior 30 days), another trial of an investigational product expected to interfere with study procedures or outcomes;
* Have breast implant(s);
* Have reconstructed breast(s).

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Balleyguier, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Lydia Liao, MD, Principal Investigator — Cooper Health; Kathy Schilling, MD, Principal Investigator — Boca Raton Regional Hospital
Locations (3):
- United States (2):
  - Boca Raton Regional Hospital Christine E. Lynn Women's Health and Wellness Institute, Boca Raton, Florida
  - Cooper Health - Cooper Breast Imaging Centers, Voorhees Township, New Jersey
- Gustave Roussy, Villejuif, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DBT and FFDM
Started | 196
Completed | 159
Not Completed | 37
Not completed — Withdrawal by Subject | 37

BASELINE CHARACTERISTICS:
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 196
Age, Customized [Count of Participants; unit: Participants]
  Age 30 years and greater | 196
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 136
  France | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DBT, FFDM and Biopsy Specimens Collected.
Description: For each participant, obtain image data using two methods (DBT and FFDM) and obtain histology results of biopsy specimens from women referred for biopsy.
Time Frame: Approximately 8 weeks
Population: Initially asymptomatic adult women presenting for breast biopsy based on prior breast imaging.
Measure: Count of Participants; unit: Participants
Groups:
- DBT and FFDM: Participants underwent 2D breast imaging with full-field digital mammography (FFDM) and by 3D breast imaging with digital breast tomosynthesis (DBT). Digital Breast Tomosynthesis: 3D imaging of the breast using Digital Breast Tomosynthesis (DBT) device. Full-Field Digital Mammography: 2D imaging of the breast using Full-Field Digital Mammography (FFDM) device.
  Subjects also were referred (per standard of care) for a biopsy. Specimen was collected, and result was recorded.
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 196
Participants
  Participants that completed DBT, FFDM and Biopsy | 159
  Participants that did not complete all three tests | 37

2. Secondary Outcome: Lesion Type Observed by FFDM Imaging
Description: Lesions were characterized based on findings identified during image evaluations performed by qualified readers.
Time Frame: Approximately 8 weeks
Population: Participants with lesions evaluated by FFDM. A single participant may have more than one lesion.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 159
Number analyzed (lesions) | 173
lesions
  Lesion description = mass | 76
  Lesion description = calcification | 67
  Lesion description = all other | 30

3. Secondary Outcome: Lesion Type Observed by DBT Imaging
Description: Lesions were characterized based on findings identified during image evaluations performed by qualified researchers.
Time Frame: Approximately 8 weeks
Population: Participants with DBT breast images collected, and lesion characteristic described by qualified reader. Participants may have more than one lesion.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 159
Number analyzed (lesions) | 192
lesions
  Lesion description = mass | 97
  Lesion description = calcification | 67
  Lesion description = all other | 28

4. Secondary Outcome: Maximum Lesion Dimension as Observed by FFDM
Description: Maximum Length of Lesions (measured in mm) when images were collected using FFDM.
Time Frame: Approximately 8 weeks
Population: Lesions observed and measured when images were collected when using FFDM; Seven (7) of the total 173 observed lesions were not measured.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: lesions
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 159
Number analyzed (lesions) | 166
millimeters (mm) | 12.45 (9.89)

5. Secondary Outcome: Maximum Lesion Dimension as Observed by DBT
Description: Maximum length of lesions (measured in mm) when images were collected using DBT
Time Frame: Approximately 8 weeks
Population: Lesions observed and measured when images were collected using DBT. Sixteen (16) of the total 192 observed lesions were not measured.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Lesions
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 159
Number analyzed (Lesions) | 176
millimeters (mm) | 12.24 (9.09)

6. Secondary Outcome: Biopsy Finding of Lesions Per Subject.
Description: Describes histologic cancer and non-cancer findings of lesion biopsy. Cancer status of lesions was reported per subject, not per lesion.
Time Frame: Approximately 8 weeks
Population: All lesions with a biopsy finding: "positive/malignant", "negative/benign" or "non-conclusive". Biopsy findings were reported per subject, not per lesion.
Measure: Number; unit: participants
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 159
participants
  Lesions identified as "positive/malignant" | 62
  Lesions identified as "negative/benign" | 94
  Biopsy was no-conclusive | 3

7. Other Pre Specified Outcome: Safety - Device Related Malfunctions
Description: Number of device-related malfunctions by imaging modality.
Time Frame: less than 16 months
Population: Number of device malfunctions recorded for either DBT or FFDM imaging.
Measure: Number; unit: malfunction events reported
Arm/Group | DBT and FFDM
Number analyzed (Participants) | 196
malfunction events reported | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from June 2015 to November 2016 (1 year and 5 months).
Arm/Group | DBT and FFDM
All-Cause Mortality (participants affected / at risk) | 0/196
Serious Adverse Events (participants affected / at risk) | 0/196
Other Adverse Events (participants affected / at risk) | 0/196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT02324205/Prot_SAP_000.pdf